CLINICAL TRIAL: NCT00761085
Title: Methadone in Pediatric and Adult Sickle Cell Patients
Acronym: MSCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201107091
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Morphine; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Methadone-Children (Active Comparator): Methadone comparison to standard of care for pain management
  Interventions: Drug: Methadone
- Morphine-Children (Active Comparator): Morphine standard of Care pain management
  Interventions: Drug: Morphine
- Methadone-Adults (Active Comparator): Methadone comparison to standard of care for pain management
  Interventions: Drug: Methadone
- Morphine-Adults (Active Comparator): Morphine standard of Care pain management
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Standard of care for pain management of acute episode of pain
  Arms: Morphine-Adults; Morphine-Children
Drug: Methadone — Compare to standard of care for pain management of acute episode of pain
  Arms: Methadone-Adults; Methadone-Children

SUMMARY:
To determine the pharmacokinetics of methadone in children and adults with SCD who are experiencing a painful episode.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 7 years and less than or equal to 40 years
* Confirmed diagnosis of any form of sickle cell disease, including sickle cell anemia, sickle-hemoglobin C disease, and sickle-B thalassemia
* Currently experiencing a vaso-occlusive episode (VOE), defined as acute pain in the extremities
* Admitted to the inpatient unit for further treatment
* Started on morphine patient controlled analgesia and infusion for pain management

Exclusion Criteria:

* Diagnosis of acute chest syndrome
* New focal neurologic findings or clinical concern of stroke
* Aplastic crisis with hemoglobin 2 g/dl below steady-state value
* Allergy to morphine or methadone
* Any other medical condition that the attending physician deems to be a contraindication to therapy
* Liver or renal insufficiency or failure, and congestive heart failure

Ages: 7 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2010-11-07 (Actual); Study Completion 2010-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan D Kharasch, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital/St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Horst J, Frei-Jones M, Deych E, Shannon W, Kharasch ED. Pharmacokinetics and analgesic effects of methadone in children and adults with sickle cell disease. Pediatr Blood Cancer. 2016 Dec;63(12):2123-2130. doi: 10.1002/pbc.26207. Epub 2016 Aug 30. PMID 27572136

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methadone-Children | Morphine-Children | Methadone-Adults | Morphine-Adults
Started | 12 | 12 | 11 | 12
Completed | 12 | 6 | 11 | 8
Not Completed | 0 | 6 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone-Children | Morphine-Children | Methadone-Adults | Morphine-Adults | Total
Number analyzed (Participants) | 12 | 12 | 11 | 12 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (2) | 14 (3) | 25 (6) | 25 (7) | 22 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 7 | 7 | 23
  Male | 8 | 7 | 4 | 5 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 11 | 12 | 47

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Pharmacokinetics of Methadone in Children and Adults With Sickle Cell Disease Experiencing a VOE.
Description: R-Methadone AUC
Time Frame: 96 hr
Measure: Mean (Standard Deviation); unit: (hr*ng/ml)
Arm/Group | Methadone-Children | Morphine-Children | Methadone-Adults | Morphine-Adults
Number analyzed (Participants) | 12 | 12 | 11 | 12
(hr*ng/ml) | 523 (248) | 0 (0) | 637 (324) | 0 (0)
Statistical Analysis 1: Comparison: Methadone-Children vs Morphine-Children vs Methadone-Adults vs Morphine-Adults; No statistical comparisons of methadone concentration in patients receiving methadone vs not receiving methadone (children or adults). No statistical comparisons of methadone concentration in children vs adults; Test type: Other — No statistical comparisons; No statistical comparisons

2. Secondary Outcome: Pain Relief
Description: Pain relief score using the 10CM VAS, which has a pain scale of 0-10, with 0=no pain and 10=worst pain experienced
Time Frame: 72 hr
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methadone-Children | Morphine-Children | Methadone-Adults | Morphine-Adults
Number analyzed (Participants) | 12 | 12 | 11 | 12
units on a scale | 8 (2) | 4 (3) | 5 (3) | 5 (2)
Statistical Analysis 1: Comparison: Methadone-Children vs Morphine-Children vs Methadone-Adults vs Morphine-Adults; Test type: Superiority; p < 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | Methadone-Children | Morphine-Children | Methadone-Adults | Morphine-Adults
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes